CLINICAL TRIAL: NCT02966678
Title: Incidence of Dyschromatopsia in Glaucoma
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Dyschromatopsia
Record Dates: First submitted 2016-11-07; First posted 2016-11-17 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Glaucoma
Keywords: Glaucoma, Dychromatopsia
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glaucoma: Patients with a diagnosis of glaucoma will undergo color vision test
  Interventions: Procedure: Color Vision Test

INTERVENTIONS:
Procedure: Color Vision Test — Farnsworth Panel D15/Hue test plus Ishihara charts

SUMMARY:
Incidence of dyschromatopsia

DETAILED DESCRIPTION:
Incidence of dyschromatopsia should be elevated in glaucoma compared to a healthy control population. However, the actual incidence rate is not investigated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of glaucoma
* age between 18 and 99 years old
* best corrected visual acuity(BCVA) > 0.2 (decimal Snellen)

Exclusion Criteria:

* age < 18 yo
* BCVA < 0.2
* known dyschromatopsia
* known corneal disease
* St.p. corneal surgeries
* macula disease
* history of medication use that can influence color vision (e.g. hydroxychloroquine)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of glaucoma from a university outpatient department
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of dyschromatopsia | first and only study visit (day 1 of the study)
  Incidence of dyschromatopsia should be elevated in glaucoma compared to a healthy control population. However, the actual incidence rate is not investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Funk, MD, PhD, Principal Investigator — UniversityHospital Zurich, Dept. of Ophthalmology

IPD SHARING:
Plan to Share IPD: No